CLINICAL TRIAL: NCT04960865
Title: Effects of Kinesio Taping on Calf Muscle Fatigue in Collegiate Female Athletes
Brief Title: Kinesio Taping and Calf Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RRC-2021-05
Record Dates: First submitted 2021-06-26; First posted 2021-07-14 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Fatigue
Keywords: Calf Muscle; Kinesio tape; Muscle fatigue; Heel raises
MeSH Terms: conditions — Fatigue | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Three-arm parallel group
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were not aware of the type of tape applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Participants will be applied Kinesio tape with 50% tension.
  Interventions: Other: Kinesio Taping under tension.
- Sham Group (Sham Comparator): Participants will be applied Kinesio tape without any tension.
  Interventions: Other: Kinesio Tape without tension
- Placebo Group (Placebo Comparator): Participants will be applied rigid tape without any tension
  Interventions: Other: Rigid Taping

INTERVENTIONS:
Other: Kinesio Taping under tension. — Kinesio tape will be applied to participants under tension.
  Arms: Experimental Group
Other: Kinesio Tape without tension — Kinesio tape will be applied to participants without any tension.
  Arms: Sham Group
Other: Rigid Taping — Rigid Taping will be applied.
  Arms: Placebo Group

SUMMARY:
Muscle fatigue results in decreased ability in muscles to generate force. Kinesio Tape may reverse the adverse effects of fatigue. Thus this study will examine the acute effects of Kinesio tape on muscle fatigue.

DETAILED DESCRIPTION:
The participants will be divided into three groups; 1. Experimental group: Kinesio tape with 50% tension will be applied; 2. Sham group: Kinesio tape without any tension will be applied; 3. Placebo group: Rigid tape without any tension will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy cooperative individuals.
* Female athletes who were engaged in training at least 3 times a week.
* The subject should perform a minimum of 23 hell raises.

Exclusion Criteria:

* Musculoskeletal injuries, cardio-pulmonary vestibular and neurological complication and systemic disorder.
* Consumption of any pre-workout supplement in the last 6 months.
* Involvement in any other training program.

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Number of heel raises | 1 week.
  Participants will have to perform heel raises in standing position untill thay are fatigued.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th., Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rana A, Tyagi D, Alghadir AH, Khan M. Effects of Kinesio taping on calf muscle fatigue in college female athletes: A randomized controlled trial. Medicine (Baltimore). 2022 Oct 28;101(43):e31004. doi: 10.1097/MD.0000000000031004. PMID 36316875